CLINICAL TRIAL: NCT05407311
Title: 64Cu-SAR-BBN Positron Emission Tomography: A Phase 2 Study of Participants With PSMA-negative Biochemical Recurrence of Prostate Cancer
Brief Title: 64Cu-SAR-BBN for Identification of Participants With Recurrence of Prostate Cancer (SABRE)
Acronym: SABRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLB03
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Biochemical Recurrence of Malignant Neoplasm of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 64Cu-SAR-BBN (Experimental): Patients will receive a single administration of 200 megabecquerels (MBq) of 64Cu-SAR-BBN.
  Interventions: Drug: 64Cu-SAR-BBN

INTERVENTIONS:
Drug: 64Cu-SAR-BBN — 64Cu-SAR-BBN

SUMMARY:
The aim of this study is to determine the safety and efficacy of 64Cu-SAR-BBN and determine the ability of 64Cu-SAR-BBN Positron emission tomography (PET)/computed tomography (CT) to correctly detect the recurrence of prostate cancer in participants with prostate-specific membrane antigen (PSMA)-negative biochemical recurrence of prostate cancer following definitive therapy.

DETAILED DESCRIPTION:
Participants with biochemical evidence of recurrence of prostate cancer (PC) were evaluated with 64Cu-SAR-BBN PET/CT (Day 0 and Day 1) and by conventional methodologies up to 180 days later (e.g., histopathology/biopsy, conventional imaging, prostate specific antigen [PSA] reduction post focal salvage therapy or radiotherapy with no concomitant androgen deprivation therapy). Three independent, central readers blinded to the participant number, the time of the PET/CT scan, and the results of the conventional methodologies, assessed the 64Cu-SAR-BBN PET/CT. Three separate independent readers assessed the results of the conventional methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Life expectancy ≥ 12 weeks as determined by the Investigator.
4. Histologically confirmed adenocarcinoma of prostate per original diagnosis and completed subsequent definitive therapy.
5. Suspected recurrence of PC based on rising PSA after definitive therapy on the basis of:

   1. Post-radical prostatectomy: Detectable or rising PSA that is ≥ 0.2 ng/mL with a confirmatory PSA ≥ 0.2 ng/mL (per American Urological Association recommendation) or
   2. Post-radiation therapy, cryotherapy, or brachytherapy: Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir (per American Society for Therapeutic Radiology and Oncology-Phoenix consensus definition).
6. Negative or equivocal findings for PC on (1) approved PSMA PET and (2) anatomical imaging (CT and/or magnetic resonance imaging) and (3) if available, any other conventional imaging performed as part of routine standard of care imaging workup within 60 days prior to Day 0.
7. The Eastern Cooperative Oncology performance status 0-2.
8. Adequate recovery from acute toxic effects of any prior therapy.
9. Estimated Glomerular Filtration Rate of 30 mL/min or higher.
10. Adequate liver function.
11. For participants who have partners of childbearing potential: Partner and/or participant must use a method of birth control with adequate barrier protection.

Exclusion Criteria:

1. Participants who received other investigational agents within 28 days prior to Day 0.
2. Participants administered any high energy (>300 kiloelectronvolts (keV)) gamma-emitting radioisotope within 5 physical half-lives prior to Day 0.
3. Ongoing treatment or treatment within 90 days of Day 0 with any systemic therapy (e.g. androgen-deprivation therapy, antiandrogen, gonadotropin-releasing hormone, luteinizing hormone-releasing hormone agonist or antagonist) for PC.
4. Participants who are known to require prohibited treatment (e.g., initiation of androgen-deprivation therapy due to rapidly rising PSA) before the 64Cu-SAR-BBN PET/CT results can be verified via histopathology or follow-up imaging.
5. Known or expected hypersensitivity to 64Cu-SAR-BBN or any of its components.
6. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Tower Urology, Los Angeles, California
  - Stanford University, Stanford, California
  - Biogenix Molecular, Miami, Florida
  - Bamf Health, Inc, Grand Rapids, Michigan
  - St Louis University Hospital, St Louis, Missouri
  - GU Research Network, Omaha, Nebraska
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period:
  19 Sep 2022 to 14 Nov 2023
Groups:
- 64Cu-SAR-BBN: Participants with suspected biochemical recurrence of prostate cancer (PC) following definitive therapy with negative or equivocal findings for PC on an approved prostate-specific membrane antigen (PSMA) positron emission tomography (PET) and anatomical imaging (computed tomography [CT] and/or magnetic resonance imaging [MRI]) and other standard of care (SOC) conventional imaging received a single intravenous injection of 200 megabecquerels (MBq) of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/-6 hours post injection.
Period: Overall Study
Arm/Group | 64Cu-SAR-BBN
Started | 53
Completed | 43
Not Completed | 10
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received any amount of 64Cu-SAR-BBN.
Groups:
- 64Cu-SAR-BBN: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53
Baseline Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 3.3932 (6.13380)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Incidence and severity of Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events. Adverse Events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: Up to 7 days post injection
Population: All Participants who received any amount of 64Cu-SAR-BBN.
Measure: Count of Participants; unit: Participants
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 53
Participants
  Any TEAE | 8
  TEAE Grade 1 to 2 | 8
  TEAE Grade 3 | 0
  TEAE Grade 4 to 5 | 0
  TEAE Related to 64Cu-SAR-BBN | 2
  Serious TEAE | 0
  TEAE Leading to Discontinuation of Study | 0
  TEAE Leading to Death | 0

2. Primary Outcome: Participant-level Correct Detection Rate (CDR) - Day 0
Description: The percentage of true positive (TP) participants on the Day 0 scan out of all participants with a Day 0 scan.
Time Frame: Day 0 (1-4 hours) post injection
Population: All participants who received any amount of 64Cu-SAR-BBN and had 64Cu-SAR-BBN PET/CT imaging results from at least one central reader, excluding participants with non-evaluable Reference Standard results or without an evaluable 64Cu-SAR-BBN PET/CT scan central reader result, at Day 0.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 47
percentage of participants
  Reader 1 | 14.9 [6.2 to 28.3]
  Reader 2 | 14.9 [6.2 to 28.3]
  Reader 3 | 14.9 [6.2 to 28.3]

3. Primary Outcome: Participant-level CDR - Day 1.
Description: The percentage of TP participants on the Day 1 scan out of all participants with a Day 1 scan.
Time Frame: Day 1 (24+/-6 Hours) post injection
Population: All participants who received any amount of 64Cu-SAR-BBN and had 64Cu-SAR-BBN PET/CT imaging results from at least one central reader, excluding participants with non-evaluable Reference Standard results or without an evaluable 64Cu-SAR-BBN PET/CT scan central reader result, at Day 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 47
percentage of participants
  Reader 1 | 4.3 [0.5 to 14.5]
  Reader 2 | 10.6 [3.5 to 23.1]
  Reader 3 | 14.9 [6.2 to 28.3]

4. Primary Outcome: Region-level Positive Predictive Value (PPV) - Day 0.
Description: The percentage of TP regions on the Day 0 scan out of all positive regions on the Day 0 scan.
Time Frame: Day 0 (1-4 hours) post injection
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of regions
Units Other Than Participants: Regions
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 47
Number analyzed (Regions) | 235
percentage of regions
  Reader 1 | 47.1 [23.0 to 72.2]
  Reader 2: number analyzed (Regions) | 219
  Reader 2 | 22.6 [9.6 to 41.1]
  Reader 3 | 33.3 [15.6 to 55.3]

5. Primary Outcome: Region-level PPV - Day 1.
Description: The percentage of TP regions on the Day 1 scan out of all positive regions on the Day 1 scan.
Time Frame: Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of regions
Units Other Than Participants: Regions
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 47
Number analyzed (Regions) | 235
percentage of regions
  Reader 1 | 22.2 [2.8 to 60.0]
  Reader 2: number analyzed (Regions) | 222
  Reader 2 | 35.3 [14.2 to 61.7]
  Reader 3 | 37.5 [18.8 to 59.4]

6. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVmean - Day 0
Description: The mean Standardized Uptake Value (SUVmean) in lesions, visceral soft tissue, bone.
Time Frame: Day 0 (1-4 hours) post injection
Population: All enrolled participants who received any amount of 64Cu-SAR-BBN who had at least one biodistribution measure. The number of participants analyzed varied depending on the number of lesions identified by each reader in each participant and in each region.
Measure: Mean (Standard Deviation); unit: kg/L
Groups:
- Reader 1; Reader 2; Reader 3: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 14 | 23 | 21
kg/L
  All Lesions | 5.470 (3.2058) | 3.773 (2.5440) | 5.671 (8.0303)
  Soft Tissue Lesions: number analyzed (Participants) | 14 | 18 | 18
  Soft Tissue Lesions | 5.699 (3.5380) | 4.362 (2.9050) | 6.427 (8.5057)
  Bone Lesions: number analyzed (Participants) | 1 | 8 | 4
  Bone Lesions | 3.703 (NA) — No standard deviation when n=1 | 2.482 (1.2925) | 2.353 (2.0118)

7. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVmean - Day 1
Description: The SUVmean in lesions, visceral soft tissue, bone.
Time Frame: Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/L
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 9 | 15 | 20
kg/L
  All Lesions | 2.586 (1.9814) | 1.450 (1.5305) | 1.179 (1.5309)
  Soft Tissue Lesions: number analyzed (Participants) | 9 | 11 | 11
  Soft Tissue Lesions | 2.586 (1.9814) | 1.586 (1.7712) | 1.652 (2.0244)
  Bone Lesions: number analyzed (Participants) | 0 | 5 | 12
  Bone Lesions |  | 2.116 (2.3684) | 0.772 (0.4263)

8. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVmax - Day 0
Description: The max Standardized Uptake Value (SUVmax) in lesions, visceral soft tissue and bone.
Time Frame: Day 0 (1-4 hours) post injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/L
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 14 | 23 | 21
kg/L
  All Lesions | 7.335 (4.0904) | 5.314 (3.1471) | 14.436 (27.7988)
  Soft Tissue Lesions: number analyzed (Participants) | 14 | 18 | 18
  Soft Tissue Lesions | 7.705 (4.7952) | 5.910 (3.8559) | 16.368 (29.7231)
  Bone Lesions: number analyzed (Participants) | 1 | 8 | 4
  Bone Lesions | 5.041 (NA) — No standard deviation when n=1 | 4.144 (1.8181) | 5.013 (3.6903)

9. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVmax - Day 1
Description: The SUVmax in lesions, visceral soft tissue and bone.
Time Frame: Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/L
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 9 | 15 | 20
kg/L
  All Lesions | 4.179 (3.3173) | 2.762 (3.5449) | 2.763 (3.2511)
  Soft Tissue Lesions: number analyzed (Participants) | 9 | 11 | 11
  Soft Tissue Lesions | 4.179 (3.3173) | 2.930 (4.1078) | 3.965 (4.5243)
  Bone Lesions: number analyzed (Participants) | 0 | 5 | 12
  Bone Lesions |  | 5.017 (6.2016) | 1.945 (0.8572)

10. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVr - Day 0
Description: Standardized Uptake Value Lesion to Background ratio (SUVr): SUVmax of the lesion divided by the SUVmean of gluteus background.
Time Frame: Day 0 (1-4 hours) post injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 14 | 23 | 21
ratio | 14.566 (8.1016) | 10.020 (5.1889) | 13.442 (17.6749)

11. Secondary Outcome: Biodistribution of 64Cu-SAR-BBN - SUVr - Day 1
Description: SUVr: SUVmax of the lesion divided by the SUVmean of gluteus background.
Time Frame: Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Reader 1 | Reader 2 | Reader 3
Number analyzed (Participants) | 9 | 15 | 20
ratio | 55.957 (36.4771) | 40.617 (24.7419) | 36.254 (45.2321)

12. Secondary Outcome: Participant-level PPV
Description: Percentage of TP participants out of all positive participants, derived separately for each timepoint and reader.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours) post injection
Population: All participants who received any amount of 64Cu-SAR-BBN and had 64Cu-SAR-BBN PET/CT imaging results from at least one central reader, excluding participants with non-evaluable Reference Standard results or without an evaluable 64Cu-SAR-BBN PET/CT scan central reader result, at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participant-level PPV - Day 0; Participant-level PPV - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Participant-level PPV - Day 0 | Participant-level PPV - Day 1
Number analyzed (Participants) | 47 | 47
percentage of participants
  Reader 1 | 58.3 [27.7 to 84.8] | 33.3 [4.3 to 77.7]
  Reader 2 | 31.8 [13.9 to 54.9] | 38.5 [13.9 to 68.4]
  Reader 3 | 36.8 [16.3 to 61.6] | 43.8 [19.8 to 70.1]

13. Secondary Outcome: Participant-level Detection Rate (DR)
Description: Percentage of participants with a positive 64Cu-SAR-BBN PET/CT scan out of all participants with a 64Cu-SAR-BBN PET/CT scan for each timepoint and reader.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours) post injection
Population: All participants who received any amount of 64Cu-SAR-BBN and had a 64Cu-SAR-BBN PET/CT scan at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participant-level DR - Day 0; Participant-level DR - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Participant-level DR - Day 0 | Participant-level DR - Day 1
Number analyzed (Participants) | 53 | 53
percentage of participants
  Reader 1 | 24.5 [13.8 to 38.3] | 17.0 [8.1 to 29.8]
  Reader 2 | 43.4 [29.8 to 57.7] | 28.3 [16.8 to 42.3]
  Reader 3 | 37.7 [24.8 to 52.1] | 37.7 [24.8 to 52.1]

14. Secondary Outcome: Participant-level False Positive Rate (FPR)
Description: Percentage of false positive (FP) participants out of all participants with a positive scan, derived separately for each timepoint and reader.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participant-level FPR - Day 0; Participant-level FPR - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Participant-level FPR - Day 0 | Participant-level FPR - Day 1
Number analyzed (Participants) | 47 | 47
percentage of participants
  Reader 1 | 41.7 [15.2 to 72.3] | 66.7 [22.3 to 95.7]
  Reader 2 | 68.2 [45.1 to 86.1] | 61.5 [31.6 to 86.1]
  Reader 3 | 63.2 [38.4 to 83.7] | 56.3 [29.9 to 80.2]

15. Secondary Outcome: Region-level FPR
Description: Percentage of FP regions on the Day 0 or Day 1 scan out of all positive regions, derived separately for each timepoint and reader.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours) post injection
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of regions
Units Other Than Participants: Regions
Groups:
- Region-level FPR - Day 0; Region-level FPR - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Region-level FPR - Day 0 | Region-level FPR - Day 1
Number analyzed (Participants) | 47 | 47
Number analyzed (Regions) | 235 | 235
percentage of regions
  Reader 1 | 52.9 [27.8 to 77.0] | 77.8 [40.0 to 97.2]
  Reader 2: number analyzed (Regions) | 219 | 222
  Reader 2 | 77.4 [58.9 to 90.4] | 64.7 [38.3 to 85.8]
  Reader 3 | 66.7 [44.7 to 84.4] | 62.5 [40.6 to 81.2]

16. Secondary Outcome: Participant-level Discrepant PET Negativity Rate
Description: Percentage of participants with contradicting Day 0 and Day 1 results for whom the Reference Standard was positive.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours) post injection
Population: All participants who received any amount of 64Cu-SAR-BBN with 64Cu-SAR-BBN PET/CT imaging results from at least one central reader and had a positive reference standard on the participant level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 64Cu-SAR-BBN
Number analyzed (Participants) | 19
percentage of participants
  Reader 1 | 26.3 [9.1 to 51.2]
  Reader 2 | 15.8 [3.4 to 39.6]
  Reader 3 | 10.5 [1.3 to 33.1]

17. Secondary Outcome: Participant-level True Negative Rate (TNR)
Description: Percentage of true negative (TN) participants on the Day 0 or Day 1 scan out of all participants with a negative Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours) post injection
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participant-level TNR - Day 0; Participant-level TNR - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Participant-level TNR - Day 0 | Participant-level TNR - Day 1
Number analyzed (Participants) | 47 | 47
percentage of participants
  Reader 1 | 82.1 [63.1 to 93.9] | 85.7 [67.3 to 96.0]
  Reader 2 | 57.1 [39.4 to 73.7] | 77.1 [59.9 to 89.6]
  Reader 3 | 58.6 [38.9 to 76.5] | 69.0 [49.2 to 84.7]

18. Secondary Outcome: Region-level TNR
Description: Percentage of TN regions on the Day 0 or Day 1 scan out of all negative regions on the Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours) post injection
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of regions
Units Other Than Participants: Regions
Groups:
- Region-level TNR - Day 0; Region-level TNR - Day 1: Participants with suspected biochemical recurrence of PC following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other SOC conventional imaging received a single intravenous injection of 200 MBq of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | Region-level TNR - Day 0 | Region-level TNR - Day 1
Number analyzed (Participants) | 47 | 47
Number analyzed (Regions) | 235 | 235
percentage of regions
  Reader 1 | 95.8 [92.2 to 98.1] | 96.7 [93.4 to 98.7]
  Reader 2: number analyzed (Regions) | 219 | 222
  Reader 2 | 88.2 [82.9 to 92.3] | 94.6 [90.6 to 97.3]
  Reader 3 | 92.6 [88.2 to 95.7] | 93.0 [88.8 to 96.0]

ADVERSE EVENTS:
Time Frame: From time of informed consent up to 7 days post injection
Description: Adverse event monitoring occurred at screening, on Day 0 pre- and post-dose, and up to 7 days post injection (Day 7). Physical exam performed pre-dose on Day 0 and on Day 7. Vital signs collected pre- and post-dose on Day 0 and on Day 7. Duplicate 12-Lead electrocardiogram (ECG) performed pre- and post-dose on Day 0. Hematology, biochemistry, coagulation, and estimated glomerular filtration rate (eGFR) performed at screening and Day 7. Urinalysis performed pre-dose on Day 0 and on Day 7.
Groups:
- 64Cu-SAR-BBN: Participants with suspected biochemical recurrence of prostate cancer (PC) following definitive therapy with negative or equivocal findings for PC on an approved PSMA PET and anatomical imaging (CT and/or MRI) and other standard of care (SOC) conventional imaging received a single intravenous injection of 200 megabecquerels (MBq) of 64Cu-SAR-BBN, followed by a PET/CT scan at 1 to 4 hours post injection and at 24 +/- 6 hours post injection.
Arm/Group | 64Cu-SAR-BBN
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 3/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 64Cu-SAR-BBN (N=53)
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may only be published by the principal investigator/institution following the first multi-site publication. The proposed publication will be submitted to Sponsor at least 90 days prior to submission to the publication to allow the Sponsor to delete Sponsor Confidential Information (other than Study results), correct any inaccuracies or delay the publication to allow for filing of patent applications.

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT05407311/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT05407311/SAP_001.pdf